CLINICAL TRIAL: NCT04594668
Title: Senicapoc in COVID-19 Patients With Severe Respiratory Insufficiency - A Randomized, Open-Label, Phase II Trial
Brief Title: Senicapoc in COVID-19 Patients With Severe Respiratory Insufficiency
Acronym: COVIPOC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001420-34
Record Dates: First submitted 2020-10-07; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-04

CONDITIONS: ARDS, Human; COVID
Keywords: senicapoc; severe acute respiratory distress syndrome; SARS-COV2; corona virus infection
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections | interventions — senicapoc

STUDY DESIGN:
Intervention Model Description: A Randomized, Open-Label, Phase II Trial
Masking Description: Senicapoc-treated patients compared to standard treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (No Intervention): Standard intensive care
- Senicapoc (Active Comparator): Senicapoc
  Interventions: Drug: Senicapoc

INTERVENTIONS:
Drug: Senicapoc — The intervention will consist of 50 mg enteral senicapoc administered as soon as possible after randomization and again after 24 hours
  Other Names: ICA-17043
  Arms: Senicapoc

SUMMARY:
SARS-CoV-2, one of a family of human coronaviruses, was initially identified in December 2019 in Wuhan city. This new coronavirus causes a disease that has now been named COVID-19. The virus has subsequently spread throughout the world and was declared a pandemic by the World Health Organisation on 11th March 2020. As of April 1, 2020, there are 874.081 numbers of confirmed cases with 43.290 fatalities. There is no approved therapy for COVID-19 and the current standard of care is supportive treatment.

Key markers implying a fatal outcome are acute respiratory distress syndrome (ARDS)-like disease with pronounced dyspnea, hypoxia and radiological changes in the lung. Senicapoc improves oxygenation and reduces fluid retention, inflammation, and bleeding in the lungs of mice with ARDS-like disease. In cells, there is an antiviral effect of senicapoc.

DETAILED DESCRIPTION:
The investigators discovered that in an animal model with a knockout of a potassium channel with intermediate conductance (KCa3.1), the knockout protected against lung damage and accumulation of liquid in the lung. In subsequent studies, the investigators have developed a mouse model showing that genetic deletion of the KCa3.1 channels and senicapoc, a blocker of KCa3.1 channels, protects against the accumulation of liquid in the lung. Moreover, senicapoc treatment possesses anti-inflammatory effects illustrated as lower leukocyte accumulation inside the lungs after injury. Importantly, it also increases the FiO2/PaO2 ratio (ratio of inhaled to blood oxygen), hence preserving lung function in mice with an ARDS-like disease. In addition, there is evidence that senicapoc has antiviral properties. Aarhus University has patented senicapoc for use in the treatment of acute respiratory disease. In this case, respiratory disease is caused by an infection with a coronavirus. Senicapoc has been developed for the treatment of sickle cell disease and has been administered to 500 patients without observation of major treatment-related adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive
* Age ≥18 years
* Respiratory insufficiency
* ICU admission

Exclusion Criteria:

* Severe heart failure (ejection fraction < 30%)
* Severe renal insufficiency (eGFR < 30 mL/min/1.73m2)
* Severe hemodynamic instability (noradrenalin dose > 0.3 μg/kg/min)
* Prior enrollment in the trial
* Pregnancy
* Allergy to senicapoc
* Inability to take enteral medication
* More than 24 hours since ICU admission
* Limitations of care
* Anticipated death within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-04-24 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | Day 3
  The PaO2/FiO2 ratio will be calculated based on the arterial gas closest to the time-point of Day 3 after randomization

SECONDARY OUTCOMES:
Ventilator-free days | Day 28
  Ventilator-free days will be defined as the number of days (or proportion of days) within the first 28 days after randomization where the patient is alive and not on invasive mechanical ventilation
Mortality | Day 28
  Assessment of mortality is considered a core outcome for trials within acute respiratory failure

OTHER OUTCOMES:
Vasopressor-free days | Day 28
  An infusion of a vasopressor will be defined as any continuous infusion of noradrenaline, dopamine, dobutamine, terlipressin, vasopressin, phenylephrine, and/or adrenaline
Sequential Organ Failure Assessment (SOFA)-score | Day 1, 2, 3, and 5
  The Sequential Organ Failure Assessment (SOFA)-score 1-4 will be used with 1 as best and 4 as worst score. The SOFA score is a validated and widely used measure of organ failure assessing the respiratory, nervous, cardiovascular, hepatic, coagulation, and renal systems. The sub scores as well as the overall SOFA score will be assessed. The calculation of the SOFA score will be based on available clinical and laboratory data. Laboratory and clinical data closest to the given time point will be used. If a given component (e.g. bilirubin) is not available, it will be assumed to be within normal ranges.
Need for renal replacement therapy | Day 28
  Renal replacement therapy includes dialysis (hemodialysis or peritoneal dialysis), hemofiltration, and hemodiafiltration.
Health-related quality of life (EQ-5D-5L) | Day 28
  Health-related quality of life (EQ-5D-5L) in 5 dimensions and 5 levels (1-5) with 1 as worst and 5 as best level in each dimension. At day 28 EQ-5D-5L will be assessed via telephone communication with the patient or a surrogate. The telephone interview will be semi-structured and based on the EQ-5D-5L questionnaire. The interview will be conducted by a centrally-located and trained member of the research team according to detailed standard operating procedures. In case the patient is still in the hospital, this interview will be face-to-face.
Measurement of SARS-CoV2 load | Day 0 and 3
  Quantification of viral load before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Christensen, MD, Principal Investigator — Aarhus University Hospital; Thomas Strøm, MD, Principal Investigator — Odense University Hospital; Bodil S Rasmussen, MD, PhD, Principal Investigator — Aalborg University Hospital; Klaus T Kristiansen, MD, Principal Investigator — Hvidovre University Hospital; Asger Granfeldt, MD, PhD, Study Chair — Aarhus University Hospital
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan: Individual de-identified participant data (including data dictionaries) will be shared following the publication of the primary and secondary endpoints as outlined in this protocol. Data to be shared included de-identified data points in published, peer-reviewed articles. Additional, related documents will also be available (study protocol, informed consent form, statistical analysis plan).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available following publication with no planned end date.
Access Criteria: Access to the data sharing will be given to researchers who provide a methodologically sound proposal for any type of analysis and requires IRB/Ethics approval (if applicable). Proposal should be addressed to us@biomed.au.dk